CLINICAL TRIAL: NCT05712213
Title: Medium Terms Outcome of sIPOM vs pIPOM in Patients Affected by Incisional Hernia
Brief Title: sIPOM vs pIPOM in Incisional Hernia Patients
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Claudio Gambardella, Clinical Professor, University of Campania Luigi Vanvitelli
Other Study IDs: sIPOM vs pIPOM
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Incisional Hernia
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pIPOM Group: Laparoscopic Incisional Hernia repair was performed with closure of fascia with non-absorbable suture (pIPOM)
  Interventions: Procedure: Intraperitoneal onlay mesh reinforcement with defect closure before placement of mesh (pIPOM)
- sIPOM Group: Laparoscopic Incisional Hernia was performed without fascia closure (sIPOM)
  Interventions: Procedure: Standard intraperitoneal onlay mesh repair (sIPOM)

INTERVENTIONS:
Procedure: Intraperitoneal onlay mesh reinforcement with defect closure before placement of mesh (pIPOM) — The pneumoperitoneum (12-15 mmHg) was built up with Veres in the Palmer'point. The primary optical trocar was set in the left upper abdomen, two other trocars were set in the left middle and lower abdomen. If necessary, adhesiolysis was firstly performed. The hernia gap was deperitonealized in order to prevent a seroma formation and, if possible, all hernia sac was removed to facilitate the healing of the hernia defect after the laparoscopic suture. This also included the transection of the ligamentum teres hepatis. We reduced the intraabdominal pressure to approx. 5 mmHg and measured the hernia gap through an intraperitoneal graduated mark. The choice of mesh size was done with an overlap of more than 5 cm. The laparoscopic closure of the hernia defect was performed with non-reabsorbable detached stitches of prolene 1/0 suture at a distance of 1.5 cm from stich to stich using a Reverdin' needle. The final fixation of the mesh took place with a non-resorbable tacks.
  Groups: pIPOM Group
Procedure: Standard intraperitoneal onlay mesh repair (sIPOM) — The pneumoperitoneum (12-15 mmHg) was built up with Veres in the Palmer'point. The primary optical trocar was set in the left upper abdomen, two other trocars were set in the left middle and lower abdomen. If necessary, adhesiolysis was firstly performed. The hernia gap was deperitonealized in order to prevent a seroma formation and, if possible, all hernia sac was removed to facilitate the healing of the hernia defect after the laparoscopic suture. This also included the transection of the ligamentum teres hepatis. We reduced the intraabdominal pressure to approx. 5 mmHg and measured the hernia gap through an intraperitoneal graduated mark. The choice of mesh size was done with an overlap of more than 5 cm. In sIPOM, the defect was not closed. The final fixation of the mesh took place with a non-resorbable tacks.
  Groups: sIPOM Group

SUMMARY:
Nowadays, two intraperitoneal mesh approaches are commonly used in Laparoscopic Ventral Hernia Repair (LVHR): the simple intraperitoneal onlay mesh repair (sIPOM) and the intraperitoneal onlay mesh reinforcement with defect closure before placement of mesh (pIPOM). The pIPOM has been introduced to reduce adverse events in incisional hernia (IH) surgery (i.e., seroma formation, recurrences etc ) associated to laparoscopic hernia repair, and satisfactory outcomes has been reported in several studies. In details, sequelae such mesh bulging seems to be less associated to pIPOM than sIPOM, even if the latter topic is matter of intense debate. The pIPOM has been introduced in the guidelines for the laparoscopic treatment of ventral and incisional abdominal wall hernias published by the International Endohernia Society (IEHS) in 2014. Despite prospective studies on the quality of IPOM-Plus are available, the evidence level for the statements in these guidelines remains low. The aim of this prospective analysis is to compare the postoperative outcomes of patients treated for Incisional hernia (IH) with sIPOM and pIPOM after 36 months follow-up in terms of recurrence and wound events.

ELIGIBILITY:
Inclusion Criteria:

* Incisional Hernia whit length >3 and <12 in width or length (Medium size according to European Hernia Society classification incisional hernias
* Body mass index (BMI) < 35 kg/m2
* Elective surgery setting
* Clean wound field according to the Centre for Disease Control and Prevention (CDC) wound classification (Grade I)

Exclusion Criteria:

* Incisional hernia <3 or >12 cm
* Abdominal aortic aneurysm disorders
* Pregnancy or lactation
* Psychiatric illness
* Multifocal hernia defect
* Life expectancy<2 years
* Inflammatory bowel disease
* emergency setting

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referring to the Departments of General Surgery of 3 Tertiary Hospitals (the "A. Rizzoli" Hospital, in Lacco Ameno Naples, the University of Campania "Luigi Vanvitelli" of Naples and the AORN "A. Cardareli" of Naples) for Incisional Hernia
Sampling Method: Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of the Hernia Recurrence (HR) postoperatively in pIPOM Group and sIPOM Group | 36 months
  Hernia Recurrence (HR) in pIPOM and sIPOM, was clinically and ultrasonographically evaluated at outpatient visit. In details, HR was clinically defined as any visible or palpable ''blowout'' in the abdominal wall. US evaluation was carried out by a radiologist with 15 years of gastrointestinal US experience. A RS85 (Samsung Madison Co Ltd., Seoul, Korea) ultrasound with a convex transducer (CA1-7A) was employed. The ultrasonic criteria of HR were a visible gap within the abdominal wall and/or ''tissue moving through the abdominal wall by Valsalva manoeuvre'' and/or a detectable ''blowout''. Size and location of all ultrasound detected HR were registered, as well as any other patient's complaint. In doubtful cases of HR, computerized tomography (CT) was performed. HR was diagnosed and recorded if clinical criteria and/or ultrasound criteria were fulfilled.
Evaluation of the Mesh Bulging (MB) rate postoperatively in pIPOM Groups and sIPOM Group | 36 months
  Mesh Bulging (MB) as any clinically evident protrusion through the hernial defect and opens into the hernial sac causing swelling. It was as well clinically and ultrasonographically evaluated at outpatient visit. US evaluation was carried out by a radiologist with 15 years of gastrointestinal US experience. A RS85 (Samsung Madison Co Ltd., Seoul, Korea) ultrasound with a convex transducer (CA1-7A) was employed. In doubtful cases of MB, computerized tomography (CT) was performed. MB was diagnosed and recorded if clinical criteria and/or ultrasound criteria were fulfilled.

SECONDARY OUTCOMES:
Evaluation of the incidence of wound events in pIPOM Group and sIPOM Group | 30 days
  The classification of wound events was assigned according to the likelihood and degree of wound contamination at the time of the operation, as stated in the Centre for Disease Control and Prevention (CDC) wound classification (superficial, deep or organ space). Surgical site events were reported according to the Ventral Hernia Working Group definitions. Actions for wound events were categorized as follows: antibiotics only, bedside wound interventions, percutaneous maneuvers or surgical debridement.
The evaluation of Quality of Life - Gastrointestinal quality of life index (GIQLI) questionnaire in pIPOM Group and sIPOM Group | 36 months
  The Gastrointestinal Quality of Life Index (GIQLI) is a validated, 36-item, self-administered questionnaire that addresses 5 domains: upper gastrointestinal symptoms (12 items), lower gastrointestinal symptoms (7 items), physical status (7 items), psychological status (5 items), and social status (5 items). Each item is quoted from 0 to 4; scores range from 0 to 144, with higher scores indicating better function. Correct or incorrect allocation was then evaluated.

REFERENCES:
- [Derived] Liang W, Liu C, Xu S, Ma S, Zong Y, Yan X. Sprint interval training for cardiovascular prevention: a time-efficient alternative or an overstated promise? An umbrella review. Eur J Appl Physiol. 2025 Sep 24. doi: 10.1007/s00421-025-05975-z. Online ahead of print. PMID 40991003
- [Derived] Pizza F, D'Antonio D, Lucido FS, Brusciano L, Mongardini FM, Dell'Isola C, Brillantino A, Docimo L, Gambardella C. IPOM plus versus IPOM standard in incisional hernia repair: results of a prospective multicenter trial. Hernia. 2023 Jun;27(3):695-704. doi: 10.1007/s10029-023-02802-2. Epub 2023 May 7. PMID 37149818